CLINICAL TRIAL: NCT07382401
Title: Developing Immersive Gamification Technology Systems For The Rehabilitation Management Of Adults With Parkinson's Disease (Phase 1 Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augmented eXperience E-health Laboratory (Other)
Collaborators: Department of Science and Technology (DOST) - Philippine Council for Health Research and Development (PCHRD) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AXEL0005
Record Dates: First submitted 2025-06-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Parkinson's Disease (PD)
Keywords: Parkinson Disease; Rehabilitation; Immersive Technology
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR-HMD (Experimental): This arm is the "VR-HMD" or virtual reality using a head-mounted display.
  Interventions: Device: VR-HMD
- AR-HMD (Experimental): This arm is the "AR-HMD" or augmented reality using a head-mounted display.
  Interventions: Device: AR-HMD
- Semi-CAVE (Experimental): This arm is the "semi-CAVE" or semi-cave automated virtual environment.
  Interventions: Device: semi-CAVE

INTERVENTIONS:
Device: VR-HMD — The immersive experience features in-game elements that can be controlled or altered upon the discretion of a therapist trained to operate the modality through a connected laptop. This modality will be used in therapy sessions administered for four sessions (twice a week for two weeks), with a maximum of 45 minutes per session. Each session would be in 10- to 20-minute periods with introduction, orientation, and provisions for rest periods for patient comfort.
  Arms: VR-HMD
Device: AR-HMD — This is similarly administered as the VR-HMD through a wearable headset. However, this modality incorporates real-world elements that support the rehabilitative exercises such as treadmills. This modality will be used in therapy sessions administered for four sessions (twice a week for two weeks), with a maximum of 45 minutes per session. Each session would be in 10- to 20-minute periods with introduction, orientation, and provisions for rest periods for patient comfort.
  Arms: AR-HMD
Device: semi-CAVE — This is administered through three short-throw projectors operated by external sensors using an outside-in tracking technology. Similar with other modalities, in-game elements can be controlled or altered upon the discretion of a therapist trained to operate the modality through a connected laptop. This modality will be used in therapy sessions administered for four sessions (twice a week for two weeks), with a maximum of 45 minutes per session. Each session would be in 10- to 20-minute periods with introduction, orientation, and provisions for rest periods for patient comfort.
  Arms: Semi-CAVE

SUMMARY:
This clinical trial aims to develop and test a prototype immersive gamification technology system (ImGTS) among healthy volunteers and to determine its acceptability, safety, and usability in a healthy population. The main question it aims to answer is:

Does ImGTS provide an acceptable, safe, and usable therapeutic modality for patients with Parkinson's Disease? Researchers will compare a head-mounted display (HMD) system and a semi cave automatic virtual environment (semi-CAVE) system to see if they are acceptable, safe, and usable as therapy for PD.

Participants will be will undergoing their assigned ImGTS intervention for four sessions (twice a week for two weeks) supervised by a trained therapist. Afterwards, they will be interviewed based on specific questionnaires used to check for acceptability, safety, and usability.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is one of the fastest growing neurological conditions worldwide. Oral medications and surgery are currently the standard of care, but these interventions are expensive and not widely available in the Philippines. Immersive technologies such as virtual reality and augmented reality applications have shown promise in improving clinical outcomes for persons with PD such as their gait and balance. However, there are currently no local immersive technology applications tailor-made for persons with PD in the Philippines. Hence, the current objective of this study is to develop and test prototype immersive gamification technology systems (ImGTS) among healthy volunteers and to determine its acceptability, safety, and usability in a healthy population. The pilot study will be divided into two stages: the development stage and the clinical trial stage. The development stage will utilize an iterative process and will involve the participation of various stakeholder groups such as caregivers of patients with PD, therapists, doctors, members of patient advocacy groups, and game development experts in order to design and develop the proposed immersive technology interventions. The clinical trial stage will utilize these prototypes and will test them among healthy volunteers for four sessions (two sessions a week for two weeks). Acceptability will be determined through the participants' responses to open ended questions on their preferences, perceptions, and experience with the ImGTS. Safety will be assessed using cybersickness questionnaires for virtual reality and augmented reality, to be supplemented with participant reports/observations of adverse events during their participation in the study. Finally, usability will be determined using the System Usability Scale, as well as through the ImGTS' performance during the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 to 70 years old
* Able to understand Filipino and English
* Montreal Cognitive Assessment - Philippines (MOCA-P) score >27
* Timed Up and Go <10 seconds

Exclusion Criteria:

* Previously diagnosed with any neurologic condition
* With any form of aphasia
* Previously diagnosed with a psychiatric disorder
* Previously diagnosed with seizures or epilepsy
* Significant visual or hearing impairment (including individuals who have difficulties seeing or hearing even with the use of assistive devices like eyeglasses or hearing aids) or use of mobility aids
* Has a history of motion sickness
* Has quadriplegia or paralysis of dominant hand
* Has a life expectancy of less than a year
* Has previously used an ImGTS (e.g., a head-mounted display (HMD) or a cave automatic virtual environment (CAVE))

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the intervention - Virtual Reality Sickness Questionnaire | Two weeks
  Safety is defined as the low or decreased incidence of adverse events with the use of the ImGTS and will be measured using the Virtual Reality Sickness Questionnaire by Kim et al., 2018 (https://doi.org/10.1016/j.apergo.2017.12.016). The questionnaire are based on the Simulator Sickness Questionnaire by Kennedy et al., 1993 (https://doi.org/10.1207/s153), and each highlight nine symptoms of cybersickness specific to VR and to AR. Symptoms are rated on a 4-point Likert scale from "None" (0) to "Severe" (3). Other adverse events observed during and after the ImGTS experience that are not covered by the questionnaires will be recorded by the researchers. Documentation of the patient's reaction and interaction with the ImGTS (including the duration of the experience, frequency of rest periods, and technical difficulties) will also be recorded by the researchers.
Safety of the intervention - Augmented Reality Sickness Questionnaire | Two weeks
  Safety is defined as the low or decreased incidence of adverse events with the use of the ImGTS and will be measured using the Augmented Reality Sickness Questionnaire by Hussain et al., 2023 (https://doi.org/10.1016/j.ergon.2023.103495). The questionnaire are based on the Simulator Sickness Questionnaire by Kennedy et al., 1993 (https://doi.org/10.1207/s153), and each highlight nine symptoms of cybersickness specific to VR and to AR. Symptoms are rated on a 4-point Likert scale from "None" (0) to "Severe" (3). Other adverse events observed during and after the ImGTS experience that are not covered by the questionnaires will be recorded by the researchers. Documentation of the patient's reaction and interaction with the ImGTS (including the duration of the experience, frequency of rest periods, and technical difficulties) will also be recorded by the researchers.
Usability of the intervention | Two weeks
  Usability is defined as the system's ability to be easy to use as determined through user perception and game performance. User perceptions will be determined using the system usability scale (SUS by Brooke, 1995). Each question has 5 response options ranging from 'Strongly agree' to 'Strongly disagree', which has a corresponding number value. Each response is added and multiplied by 2.5 to obtain the final score that ranges from 0 to 100. A SUS score above 68 is considered above average. The SUS will be used after each session and will require about 10 minutes to complete. More specific metrics on the system's performance, including an assessment of the environmental factors of usability, will also be developed once the game itself has been made. These metrics will be based on input from the researchers and the stakeholders during the FGD(s) of the pilot studies.
Acceptability of the intervention | Two weeks
  Acceptability is defined as the positive perceptions toward the ImGTS as a game and as a therapeutic tool, which will be assessed using open-ended questions. Participants during the ImGTS development stage will be asked these questions during an FGD, while the healthy volunteers (non-stakeholders) during the clinical trial will be interviewed (semi-structured) after completing each session. Questions on specific game components will be added for the clinical trial once the prototype development has been completed.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Dominic G Jamora, MD, PhD, Principal Investigator — University of the Philippines Manila
Locations (1):
- Augmented Experience eHealth Laboratory, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The website is the official website of the laboratory — https://axel.upm.edu.ph